CLINICAL TRIAL: NCT03247335
Title: Follow-up of Arthrosurface HemiCAP Implants
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Arthrosurface, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-341
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Follow-up of Arthrosurface HemiCAP shoulder implants.

DETAILED DESCRIPTION:
In summary, the investigators would like to contact all patients who have had HemiCAP implants done at CCF with at least 2 years of follow-up after their procedure. The investigators will use electronic or written means to alert the patients that they will be contacted by our team to discuss their surgery and any related issues. Once the appropriate consent is obtained, the investigators will use a brief telephone interview to ask the patients several questions regarding any re-operations or complications the patients have had since the index procedure.

ELIGIBILITY:
Inclusion Criteria:

-Patients who had Arthrosurface (Franlin, MA) HemiCAP implants placed into their shoulders at the Cleveland Clinic

Exclusion Criteria:

* Anyone who has not had ARthrosurface (Franlin, MA) HeiCAP implants placed into their shoulders at the Cleveland Clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had Arthrosurface (Franlin, MA) HemiCAP implants placed into their shoulders at the Cleveland Clinic
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Arthrosurface | 2 year
  survival curve for the implant

SECONDARY OUTCOMES:
Rate of revision surgeries | 2 year
  rate of revision surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Spindler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No